CLINICAL TRIAL: NCT01692470
Title: A Post-Marketing Surveillance Study on the Safety and Effectiveness of Rilpivirine Hydrochloride Among Adult Filipino Patients With Human Immunodeficiency Virus Type-I Infection
Brief Title: A Study on the Safety and Effectiveness of Rilpivirine Hydrochloride (Edurant) Among Adult Filipino Patients With Human Immunodeficiency Virus Type-I Infection
Status: Withdrawn | Type: Observational
Why Stopped: The company decided to cancel this study in conformity with Philippines FDA Circular 2013-004
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100849; TMC278IFD4002 (Other: Janssen Pharmaceutica); EDUPHLMA1 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Human Immunodeficiency Virus Type 1 (HIV-1) Infection
Keywords: Human immunodeficiency virus type 1 (HIV-1) infection; HIV-1; Anti-retroviral naive; ARV; Filipino patients; Rilpivirine hydrochloride; Edurant
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — Rilpivirine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- rilpivirine hydrochloride: Patients will be taking 1 tablet of 25 mg rilpivirine hydrochloride is administered once daily orally in combination with other anti-retroviral (ARV) medications.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — Patients will be taking rilpivirine hydrochloride as per the dosing regimen given on product insert approved in Philippines (ie, 1 tablet of 25 mg orally once a day) in combination with anti-retroviral (ARV) medications.
  Other Names: Edurant

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of rilpivirine hydrochloride in combination with other anti-retroviral (ARV) medications for the treatment of ARV-naive (patients who have not been exposed to ARV) Filipino patients with human immunodeficiency virus type 1 (HIV-1) infection.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the study medication), multi-center, observational (study in which the investigators/ physicians observe the patients and measure their outcomes) study. The total duration of the study will be 3 years, and approximately 60 patients who would use rilpivirine hydrochloride in routine clinical practice with a dosing regimen stipulated in the product insert (ie, 25 mg once a day) will be enrolled. As this is an observational study, assessment of patients will be based on the accepted clinical practice in the Philippines. Patients will be monitored from baseline and throughout the 48-week (2nd, 4th, 8th, 12th, 24th, 36th and 48th weeks) treatment period of rilpivirine hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Filipino patients
* ARV naive patients with HIV-1 infection who are assessed by the physician to be eligible for treatment with ARVs
* Patients who voluntarily signed the informed consent form

Exclusion Criteria:

* Patients receiving drugs known to prolong QTc intervals, medicinal products with a known risk of Torsade de Pointes and anticonvulsants, systemic dexamethasone, proton pump inhibitors
* Any previous treatment for HIV
* Previously documented HIV-2 infection
* Patients with viral load of >100,000 HIV-1 ribo nucleic acid (RNA) copies/ml
* Severely ill patients like those with acute acquired immune deficiency syndrome (AIDS)-defining illness or other major concomitant - disease prior to enrolment
* Patients with severe hepatic impairment
* Known hypersensitivity to rilpivirine hydrochloride
* Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino anti-retroviral (ARV) naive patients with human immunodeficiency virus type 1 (HIV-1) infection and who are using rilpivirine upon its local registration
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incidence of adverse events | From the date of first exposure of study medication until 30 days after the last exposure of the patient to the study medication, as assessed for 3 years
Number of patients with incidence of discontinuation of study medication due to adverse events | From the date of first exposure of study medication until 30 days after the last exposure of the patient to the study medication, as assessed for 3 years

SECONDARY OUTCOMES:
Number of patients who will not experience death due to acquired immune deficiency syndrome (AIDS) related events occurring after 6 months of treatment | Week 24, 36 and 48
Number of patients who will not develop virologic failure | Baseline (Week 1), Week 8, Week 24 and Week 48
  Virologic failure defined as a persistently detectable viral load in a patient with previously suppressed human immunodeficiency virus ribo nucleic acid (HIV RNA) or the inability to achieve an undetectable viral load after 24 weeks of therapy. The level of undetectable load is less than 50 HIV-1 RNA copies/ml.
Number of patients who will not develop immunologic failure | Baseline (Week 1), Week 24 and Week 48
  Immunologic failure defined as either of the following conditions: a) CD4 count below 100 cells/mm3 after 6 months of therapy; b) return to or a fall below, the pre-therapy CD4 baseline after 6 months of therapy; c) a 50% decline from the on-treatment peak CD4 value (if known)
Number of patients who will not have emergence of new (ie, not present at baseline) AIDS defining conditions while on treatment | Baseline (Week 1), Week 2, 4, 8, 12, 24, 36 and 48
  AIDS defining conditions may include: HIV wasting syndrome, pneumocystis jiroveci, recurrent severe bacterial pneumonia, chronic herpes simplex infection, esophageal candidiasis, extrapulmonary tuberculosis etc.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica